CLINICAL TRIAL: NCT07309796
Title: The Effect of Strengthening Exercises for Humeral Head Depressor Muscles on Clinical Outcomes After Reverse Shoulder Arthroplasty
Brief Title: Strengthening Exercises for Humeral Head Depressor Muscles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20251224
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Reverse Shoulder Arthroplasty; Depressor Muscle Training; Shoulder Rehabilitation
Keywords: Reverse shoulder arthroplasty; Depressor muscle training. Shoulder; Arthroplasty

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation Group (Active Comparator): Participants undergoing reverse shoulder arthroplasty will receive a standard conventional rehabilitation program starting at postoperative 6 th week . The patient will receive treatment 5 days a week for 6 weeks, for a total of 30 sessions. The program consists of passive, active-assisted, and active/resisted exercises.
  Exercises Included:
  Passive / Assisted
  * Scapular mobilization
  * Scapular clock
  * Passive external rotation with a stick Passive → Active-Assisted
  * Active-assisted flexion and abduction with a stick
  * Glenohumeral joint mobilization Active / Light Resistance
  * Scapular retraction
  * Light-resistance strengthening of biceps, triceps, and serratus anterior using a theraband Active / Resistance
  * Theraband-based resisted biceps, triceps, and serratus anterior strengthening
  * Continuation of glenohumeral mobilization
  * Flexion and abduction above 90°
  * Posterior capsule stretching
  Interventions: Other: Conventional Rehabilitation Group
- Depressor Muscle Strengthening Program (Experimental): Participants will receive specific strengthening exercises targeting the shoulder depressor muscles in addition to the conventional rehabilitation program. These exercises will be performed throughout the 6-week intervention period.
  Additional Exercises:
  Latissimus dorsi: Seated rowing exercise - 3 sets × 10 repetitions Pectoralis major: Supine fly exercise - 3 sets × 10 repetitions Teres major: Prone shoulder adduction, extension, and internal rotation exercise
  Interventions: Other: Conventional Rehabilitation Group; Other: Depressor Muscle Strengthening Group

INTERVENTIONS:
Other: Conventional Rehabilitation Group — After randomization and baseline assessments, participants will undergo a standard 6-week postoperative shoulder rehabilitation program, consisting of range-of-motion exercises, scapular stabilization training, and progressive strengthening. No additional depressor muscle-specific exercises will be applied.
Other: Depressor Muscle Strengthening Group — After randomization and baseline assessments, participants will receive a 6-week rehabilitation program consisting of conventional postoperative shoulder rehabilitation combined with a specific strengthening protocol targeting the shoulder depressor muscles.
  Arms: Depressor Muscle Strengthening Program

SUMMARY:
Postoperative rehabilitation after reverse shoulder arthroplasty aims to improve pain control, range of motion, and functional capacity. However, studies examining the effects of strengthening exercises targeting the humeral head depressor muscles are limited. This randomized controlled trial will evaluate the effects of adding a specific strengthening program to standard rehabilitation on pain, range of motion, quality of life, and functional outcomes.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty (RSA) is an effective surgical method, particularly in cases of massive rotator cuff tears that lead to irreversible loss of shoulder function. The primary goals of postoperative rehabilitation are to reduce pain, improve shoulder joint functions, optimize scapulothoracic rhythm, and safely restore functional use. However, studies examining the effects of specific strengthening exercises targeting the humeral head depressor muscle group (latissimus dorsi, teres major, infraspinatus, etc.) on clinical outcomes are quite limited. This study aims to evaluate the effects of a specific strengthening protocol designed for the humeral head depressor muscles following reverse shoulder arthroplasty on pain, range of motion (ROM), quality of life, functional status, and psychological well-being. Planned as a randomized controlled trial, the research will apply an additional humeral head depressor muscle strengthening program to the standard conventional rehabilitation protocol in the experimental group, while the control group will receive only the standard rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary reverse total shoulder arthroplasty Intact teres minor confirmed by physical examination (Hornblower's test) and intraoperative assessment Ability to participate in physiotherapy or a home exercise program

Exclusion Criteria:

* Active infection Deltoid muscle insufficiency Inability or unwillingness to comply with randomization Prior shoulder arthroplasty on the same side Unwillingness to participate Inability to read or understand written instructions

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analog Scale - VAS) | 6 weeks
  Pain intensity will be assessed using the Visual Analog Scale, a 10-cm line ranging from "no pain" to "worst imaginable pain." The distance from the "no pain" anchor to the participant's mark will be measured in millimeters (0-100 mm), with higher scores indicating higher pain intensity.
Upper Extremity Disability (Disabilities of the Arm, Shoulder and Hand Questionnaire - DASH) | 6 weeks
  The DASH is a 30-item self-administered questionnaire assessing upper-extremity functional limitations. Items are scored 1-5 and converted to a 0-100 scale, where higher scores indicate greater disability.
Shoulder Range of Motion (ROM) | 6 weeks
  Active shoulder flexion, abduction, external rotation, and internal rotation will be measured using a standard goniometer. Results will be recorded in degrees (°).

SECONDARY OUTCOMES:
Shoulder Function (American Shoulder and Elbow Surgeons Score - ASES) | 6 weeks
  The ASES score includes pain and functional assessments, yielding a total score between 0 and 100. Higher scores represent better shoulder function.
Thoracic Kyphosis Angle (Spinal Mouse Assessment) | 6 weeks
  Thoracic spine curvature will be evaluated using the Spinal Mouse device during flexion and extension. The system provides non-invasive, objective measurements of thoracic kyphosis.
Pain Catastrophizing (Pain Catastrophizing Scale - PCS) | 6 weeks
  The PCS consists of 13 items assessing rumination, magnification, and helplessness. Total scores range from 0 to 52, with higher scores indicating greater catastrophizing.
Anxiety and Depression (Hospital Anxiety and Depression Scale - HADS) | 6 weeks
  HADS includes 14 items (7 anxiety, 7 depression), each scored 0-3. Higher scores indicate higher levels of anxiety or depression.
Kinesiophobia (Tampa Scale of Kinesiophobia - TSK) | 6 weeks
  The TSK is a 17-item tool measuring fear of movement and reinjury. Scores range between 17 and 68, with higher scores indicating greater kinesiophobia.
Quality of Life (12-Item Short-Form Health Survey - SF-12) | 6 weeks
  The SF-12 generates Physical Component Summary (PCS) and Mental Component Summary (MCS) scores ranging from 0 to 100. Higher scores reflect better health-related quality of life.